CLINICAL TRIAL: NCT04150432
Title: Propofol in Expiratory Air, a Comparison With Plasma Propofol, BIS Value and Calculated Plasma Concentration During General Anesthesia in Children
Brief Title: Correlation Between Exhaled Propofol Concentration With Plasma Concentration in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Johan C Ræder, Professor, Consultant, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Exhaled propofol Children
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Intervention Model Description: Consecutive patients will participate in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- propofol (Experimental): propofol general anesthesia, exhaled measurement of propofol
  Interventions: Device: Edmon

INTERVENTIONS:
Device: Edmon — New device for exhaled propofol concentration measurements

SUMMARY:
Children due for elective eye surgery in propofol based anesthesia will be kept at steady state propofol infusion for maintenance, ventilation via endotracheal tube. Exhaled propofol will be measured continously by Edmon (R) (BBraun) monitor and compared with arterial plasma samples of propofol, drawn 3-5 times during the procedure.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the correlation between simultaneous concentrations of propofol in plasma and expiratory air in children during general anesthesia.

Key secondary objectives include correlating plasma and exhaled measurements of propofol with electroencephalogram (BIS) values and computer estimated propofol concentrations in plasma and brain (TCI: target control infusion) Primary endpoint: Exhaled air and plasma concentration ratios of propofol during general anesthesia in children.

ELIGIBILITY:
Inclusion Criteria:

* elective eye surgey

Exclusion Criteria:

* known propofol hypersensitivity

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Propofol plasma concentration versus simultaneous exhaled concentration | 5 hours
  repeated blood samples of propofol concentration

SECONDARY OUTCOMES:
Propofol exhaled correlation versus Bispectral Index value (BIS) | 5 hours
  repeated blood samples of propofol concentration

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Thagaard, MD, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No